CLINICAL TRIAL: NCT01829789
Title: Group Community Reinforcement Training for Parents of Treatment-Elusive Youth
Brief Title: Individual vs. Group Community Reinforcement Training to Help Parents of Substance-using Treatment-refusing Youth
Acronym: POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA034301 (NIH)
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Substance Use Disorders; Treatment Refusal
Keywords: Adolescents; Teens; Parents; Parenting; Substance Abuse; Treatment Efficacy
MeSH Terms: conditions — Substance-Related Disorders; Treatment Refusal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-CRT (Experimental): Group Community Reinforcement Training for parents
  Interventions: Behavioral: Group Community Reinforcement Training for Parents
- I-CRT (Active Comparator): Individual Community Reinforcement Training for parents
  Interventions: Behavioral: Individual Community Reinforcement Training for Parents

INTERVENTIONS:
Behavioral: Group Community Reinforcement Training for Parents
  Other Names: G-CRT
  Arms: G-CRT
Behavioral: Individual Community Reinforcement Training for Parents
  Other Names: I-CRT
  Arms: I-CRT

SUMMARY:
The purpose of this study is to test the efficacy and cost-effectiveness of Community Reinforcement Training (CRT) provided in a group therapy format. The goals of CRT are to teach parents behavioral and communication skills to influence their youth's drug use and encourage them to enter treatment. Thirty parents will be randomly assigned to Group CRT and 30 will be randomly assigned to traditional, Individual CRT. Youth engaged in treatment will receive individual Cognitive Behavioral Therapy. Families are assessed for adolescent substance use and other areas of individual and family functioning. It is expected that Group CRT will be more effective for encouraging youth entry into treatment and improving parental functioning.

DETAILED DESCRIPTION:
Very few youth with drug abuse or dependence in the United States receive treatment. This population of untreated youth represents a massive "treatment gap" in adolescent health care that renders impotent a potentially important avenue for preventing chronic drug abuse and related difficulties. The lack of motivation for treatment characterizing most adolescent drug abusers significantly decreases the likelihood these youth will enter treatment, barring mandates from the legal system or other social institutions. Efficacy studies have demonstrated that Community Reinforcement Training (CRT), an approach that involves teaching parents how to engage their youth into treatment, can work to recruit 60-80% of these treatment-elusive youth. CRT is traditionally provided in an individual therapy format to one or both parents. This study will improve upon our prior work by using a group format to provide a less costly procedure for engaging youth into treatment and to make it more portable to treatment agencies, schools, juvenile justice, and other community organizations seeking to offer support to parents or engage youth in treatment, thus significantly increasing the adoption and sustainability of the approach.

This study will examine the efficacy of the group format (G-CRT) for helping parents engage their unmotivated, resistant youth in treatment compared to the traditional individual format (I-CRT). Parents (n = 60) will be randomly assigned to G-CRT or to I-CRT. We will evaluate the differential efficacy of G-CRT, relative to I-CRT, on rates of adolescent engagement in treatment. We expect that G-CRT, compared to I-CRT, will also be associated with greater parent encouragement of adolescent sobriety, perceived social support, and family functioning. We also predict that changes on these process variables will predict increased success in engaging adolescents. We will also examine treatment outcomes for youth engaged in Cognitive Behavioral Therapy as a function of parental involvement in G-CRT or I-CRT. We predict enhanced support received by parents in G-CRT will result in greater reductions in drug use and lower levels of HIV-risk behaviors, outcomes hypothesized to be mediated by motivation to change and sessions attendance. Finally, we will conduct an informal cost-effectiveness analysis to derive preliminary estimates of the relative costs of each treatment modality per outcome unit and hypothesize that G-CRT will be more cost effective than I-CRT by virtue of having higher clinical effectiveness and lower costs. Successful outcomes here will provide the basis for a full clinical trial with larger samples.

ELIGIBILITY:
Inclusion Criteria:

* Parents have an adolescent between 15-20 years
* Parents have had contact with the adolescent on at least 40% of the past 12 weeks
* Parents have some knowledge or evidence that the adolescent would meet DSM-IV diagnostic criteria for a substance use disorder
* Adolescent has explicitly refused to attend any intake or therapy sessions
* Adolescent is not under a current court mandate for treatment or has refused to comply with the mandate
* English-speaking capability (parents and adolescents)

Exclusion Criteria:

* Evidence of adolescent psychotic or organic state of sufficient severity to interfere with understanding of study instruments and procedures
* Adolescent had received drug treatment (except detoxification) in the past 12 weeks.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Adolescent treatment engagement | 4 months
  An adolescent may enter the CBT treatment program ("treatment engagement") at any point during the 4-month time period after his or her parents begin I-CRT or G-CRT therapy.

SECONDARY OUTCOMES:
Timeline Followback (TLFB) interview | 9 months
  The TLFB is an interview to assess the quantity, frequency, and pattern of illicit substance use. Parents provide collateral data on their adolescents' substance use in the 3 months prior to enrollment. Adolescents report on their own substance use for the 3 months prior to their parents' enrollment through 6 months after enrollment.

OTHER OUTCOMES:
Medical Outcome Studies Social Support Survey | 9 months
  The MOS consists of four support subscales (Emotional/Informational, Tangible, Affectionate, and Positive Social) and an overall functional social support index. This measure will be completed by parents at baseline (about the 3 months prior to enrollment) and at 3- and 6-month follow-up points. It will be used to compare perceived social support for parents in the G-CRT versus I-CRT interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Erica M Finstad, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Center for Family and Adolescent Research, Portland, Oregon, United States